CLINICAL TRIAL: NCT06493773
Title: Alcohol Misuse Treatment Delivered in the Hepatology Clinic to Patients Newly Diagnosed With Alcohol-related Liver Disease: a Randomized Controlled Trial
Brief Title: Alcohol Misuse Treatment to Patients Newly Diagnosed With Alcohol-related Liver Disease: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Center for Clinical Research and Prevention (Network); Novavi Outpatient Clinics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SJ-895
Record Dates: First submitted 2024-06-28; First posted 2024-07-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Liver Diseases, Alcoholic; Alcohol Use Disorder; Treatment Adherence; Alcoholism; Liver Disease; Alcohol-Related
Keywords: Alcoholic liver disease; Alcohol use disorder; Alcohol treatment; randomized clinical trial; hepatology clinic
MeSH Terms: conditions — Liver Diseases, Alcoholic; Alcoholism; Treatment Adherence and Compliance; Liver Diseases | interventions — Ethanol

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: There is follow-up for each individual participant conducted by personnel blinded to the randomization and consisting of: 1) telephone contact with interview about alcohol consumption using the time-line follow-back method conducted at three time points after 1, 3 and 6 months, 2) measurement of phosphatidyl ethanol after 6 months, and 3) electronic health records from hospital and alcohol treatment facility after 6 months.
  Use of hypothesis blinding for patients about the study aim. Usual care providers in the hospital such as physicians and nurses will not see any description of AUD treatment in the medical charts.
  Analyses will be performed in a blinded data set with treatment allocation labeled "A" and "B". Prior to this, the statistical analysis plan will be completed, signed, and uploaded at clinicaltrials.gov, and the data set will be locked. Unblinding will not occur until all analyses are performed (expected autumn 2028).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care group (No Intervention): Patients randomized to standard care will receive standard supporting care by their care providers, entailing education on the nature of alcohol-related liver disease and encouragement to abstain from alcohol use.
- Intervention group (Experimental): Patients randomized to the intervention group.
  Interventions: Behavioral: Offer of specialized alcohol use disorder treatment in the hepatology clinic

INTERVENTIONS:
Behavioral: Offer of specialized alcohol use disorder treatment in the hepatology clinic — Patients are offered specialized alcohol use disorder treatment in the hepatology clinic by an experienced AUD therapist from the AUD facility. Also medical AUD treatments will be offered to support abstinence.
  Arms: Intervention group

SUMMARY:
To evaluate the efficacy of systematically offering newly diagnosed ALD patients to AUD treatment, in the hepatology clinic, on alcohol abstinence after 6 months. The investigators will conduct a randomized controlled superiority trial with parallel group design, hypothesis blinding and blinded outcome assessment comparing A) a offer to specialized AUD treatment (intervention) and B) standard care (control). Existing observational cohort ALD members will contribute to the control group in addition to the randomized controls. The primary outcome is abstinence throughout the last 30 days assessed 6 months after randomization.

DETAILED DESCRIPTION:
The investigators have designed a randomized controlled superiority trial to investigate the effectiveness of systematically offering AUD treatment in the hepatology clinic to newly diagnosed ALD patients to increase the proportion that are abstaining from alcohol after 6 months compared to standard care. The study will be embedded in an existing observational cohort from which already included participants will be used as controls in the RCT (n = 89). Please see Figure 1 for the flow of participants in the study. From november, 2025, the investigators will start to randomize eligible participants.

Randomization will take place in connection with the first visit in the observational cohort study. Study participants randomized as controls will receive standard care through their treating physicians, which consists of individualized education on the nature of ALD as well as encouragement of alcohol use cessation.

Patients in the intervention group will receive standard care in addition to an offer of AUD treatment in the hepatology clinic.

ELIGIBILITY:
Inclusion criteria

* Age > 18 years
* Newly diagnosed alcohol-related liver disease, defined as within six months from baseline visit.
* A liver stiffness above 8.0 kPa with 10 successful measurements and an interquartile range of less than 30% as assessed with transient elastography.
* Excessive alcohol consumption defined as >7 units/week for women and >14 units/week for men within the previous year.
* The patient is able to understand the purpose of the study and give informed oral and written consent to participate.

Exclusion criteria

* Not enough proficiency in Danish to participate in interviews and questionnaires.
* Pregnancy
* Ongoing specialized AUD treatment. Self-help groups and AUD counselling at general practitioners are not counting as specialized AUD treatment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported alcohol abstinence in the last 30 days at 6 months followup in combination with phosphatidylethanol level at 6 months | 6 months after baseline
  Self-reported alcohol abstinence (defined as zero consumption of alcohol) throughout the last 30 days assessed after 6 months assessed by the timeline followback method (questionnaire) and review of medical charts and measurement of phosphatidylethanol at 6 months

SECONDARY OUTCOMES:
Self-reported alcohol abstinence in the last 30 days at 3 months followup | 3 months after baseline
  Self-reported alcohol abstinence (defined as zero consumption of alcohol) throughout the last 30 days assessed after 3 months and no indications of alcohol use in medical charts.
Rate of AUD treatment | 6 and 12 months after baseline
  Any treatment for alcohol use disorder after 6 and 12 months
Rate of individuel AUD treatment | 6 and 12 months after baseline
  Any individuel treatment for alcohol use disorder after 6 and 12 months
Rate of AUD treatment | 6 and 12 months from baseline
  Number of received sessions of treatment for alcohol use disorder after 6 and 12 months
Reduction in drinks per week | 3, 6 and 12 months from baseline
  Reduction in drinks per week after 3, 6 and 12 months compared to baseline (yes or no)
Reduction in phosphatidylethanol | 6 and 12 months from baseline
  Reduction in phosphatidylethanol value at 6 and 12 months compared to baseline (yes or no)
Complications from liver disease | 3 years from baseline
  Time to first decompensation event, which is defined as variceal haemorrhage, ascites grade 2 or worse, or hepatic encephalopathy West-Haven grade 2 or worse
All-cause mortality | 3 years from baseline
  time to death
Progression of liver disease | 3 years from baseline
  Progression in liver fibrosis grade assessed by transient elastography or progression to a worse Child-Pugh class (A to B or C and B to C
Duration of AUD treatment | 6 and 12 months from baseline
  Duration of AUD treatment
Group AUD treatment sessions | 6 and 12 months from baseline
  Amount of group AUD treatment sessions
Self-reported abstinence last 30 days after 12 months and phosphatidylethanol level after 12 months | 12 months
  Self-reported alcohol abstinence last 30 days by 12 months assessed by the timeline followback method (questionnaire) and review of electronic medical records in combination with measured phosphatidylethanol level.

CONTACTS AND LOCATIONS:
Overall Officials: Lone G Madsen, PhD, Study Chair — Zealand University Hospital, Koege
Locations (1):
- Department of Medicine, Zealand University Hospital, Køge, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No
Because of the relatively low number of patients, data are considered highly sensitive and cannot allow sharing

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT06493773/Prot_SAP_000.pdf